CLINICAL TRIAL: NCT00646789
Title: A Multicenter, Open-Label, Single Dose Study to Evaluate the Safety, Tolerability and Plasma Concentration Profiles of MK0633 in Asthmatic Children Aged 12 to Less Than 16 Years
Brief Title: A Study to Evaluate the Safety, Tolerability and Plasma Concentration Profiles of MK0633 in Asthmatic Children Aged 12 to Less Than 16 Years (0633-019)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0633-019; MK0633-019; 2008_514
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

ARMS (1):
- 1 (Experimental): MK0633
  Interventions: Drug: Comparator: MK0633

INTERVENTIONS:
Drug: Comparator: MK0633 — patients will receive single 50mg oral dose with follow-up observation for 5 weeks.

SUMMARY:
To evaluate the safety, tolerability and pharmacokinetics (PK) of MK0633 in adolescent mild-to-moderate asthma patients to permit further clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

* Patient is judged to be in good health, other than having mild to moderate asthma, based on medical history, physical examination, vital signs, and laboratory safety tests
* Patient has no clinically significant abnormality on electrocardiogram (ECG) performed at the prestudy (screening) visit and/or prior to administration of the initial dose of study drug
* Patient has at least 1 year of mild-to-moderate asthma
* Patient has been a nonsmoker for at least 6 months
* Patients of childbearing potential must agree to use a medically acceptable method of contraception during the study and for 90 days after the last dose of study drug
* Patients must be able to swallow tablets

Exclusion Criteria:

* Patient has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, other than asthma, or genitourinary abnormalities or diseases
* Patient has required a visit to a hospital or emergency room due to an asthma exacerbation within 3 months of the prestudy visit
* Patient has unresolved signs and symptoms of an upper respiratory tract infection (URI) or has had had an upper respiratory tract infection within 3 weeks prior to the prestudy visit
* Patient has a history of stroke, chronic seizures, or major neurological disorder
* Patient has a history of neoplastic disease
* Use of theophylline, Singulair (montelukast), Xolair (omalizumab), Zyflo amd Zyflo CR (zileuton), oral corticosteroids and oral beta agonists are excluded approximately 2 weeks prior to administration of study drug and throughout the study
* Patient consumes alcoholic beverages

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of MK0633 in adolescent asthma patients. | Blood and urine samples will be collected at specified intervals for 72 hours after study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC